CLINICAL TRIAL: NCT03893318
Title: Intravenous Lidocaine to Reduce Postoperative Opioid Consumption and Improve Recovery After Posterior Spinal Fusion for Adolescent Idiopathic Scoliosis
Brief Title: IV Lidocaine in Pediatric AIS
Acronym: PEDS LIDO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI moved to a different institution.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201807071
Record Dates: First submitted 2019-02-21; First posted 2019-03-28 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Systemic Lidocaine Improves Pain Control After Surgery by Attenuating the Systemic Inflammatory Response to Surgery
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: a randomized, triple-blind, placebo-controlled trial of intravenous lidocaine in the management of surgery performed for adolescent idiopathic scoliosis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study Drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Group (Experimental): will receive intravenous lidocaine during and after posterior spinal fusion for AIS
  Interventions: Drug: IV lidocaine
- Control Group (Placebo Comparator): will receive saline placebo during and after surgery.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: IV lidocaine — an amide-type, short-acting local anesthetic and delivered as an aqueous solution for intravenous administration. It has a half-life of 1.5-2 hours. A traditional method of administration is via epidural delivery. Epidural lidocaine is effective and this effect is due, in part, to systemic absorption. Systemic (intravenous) administration of lidocaine is a Food and Drug Administration approved method of delivery. Low plasma levels are needed for effective use, 0.5µg/mL to 5.0µg/mL. Given this low concentration required and the short half-life, continuous infusion of lidocaine is thought to be generally safe with low risk of complication.
  Arms: Study Group
Drug: Placebos — Saline
  Arms: Control Group

SUMMARY:
This study addresses the focus areas of Post-Operative Pain Management. We propose a randomized, triple-blind, placebo-controlled trial to investigate the efficacy of a systemic infusion of intravenous lidocaine as a non-opioid method of post-operative pain management following postoperative spinal fusion for adolescent idiopathic scoliosis (AIS). The outcomes assessed will be (1) the effect of intravenous lidocaine on post-operative opioid consumption, both in-hospital and at three-month follow-up, (2) the effect of intravenous lidocaine on the immunophenotype expressed following surgery, and (3) the effect of intravenous lidocaine on recovery from surgery as assessed by the Patient Reported Outcomes Measurement Information System-Computer Adaptive Tests for Pain Interference (PI) and Mobility (M) (PROMIS-CAT). Thus, we propose a study of a non-opioid method of pain control to minimize opioid consumption in-hospital and at three-months postoperatively, with primary outcomes measures that include morphine-equivalent opioid consumption and PROMIS-Mobility to assess recovery. In addition, we will test the ability of systemic lidocaine to attenuate the systemic inflammatory response to major spine surgery. The immunologic response to surgery has been associated with rehabilitation and recovery following total hip arthroplasty and this study will provide data to support further work.

DETAILED DESCRIPTION:
a Phase IV, randomized, triple-blind, placebo-controlled trial with two study groups: postoperative standard of care with opioid patient controlled analgesia (PCA) and IV lidocaine infusion versus postoperative standard of care plus normal saline placebo. Block randomization into one of the two groups will be based on a random table generated using an R-program. Group 1 (Study) will receive intravenous lidocaine during and after posterior spinal fusion for AIS. Group 2 (Control) will receive saline placebo during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent idiopathic scoliosis indicated for posterior spinal fusion.
2. Ages between 12 and 18 years of age.
3. Parent/Guardian capable of providing informed consent for study participation

Exclusion Criteria:

1. Age < 12 or > 18 years old.
2. Unable to obtain consent for the surgical intervention or study, or if mental capacity prohibits the ability to provide consent and complete patient-reported outcomes tools.
3. Diagnosis of sepsis or infection
4. Diagnosis of primary or metastatic malignancy.
5. Participation in another clinical trial.
6. Past or current diagnoses of a cardiac arrhythmia or first/second degree heart block.
7. Past or current seizure disorders.
8. Allergy to bupivacaine.
9. Planned anterior approaches for treatment of scoliosis deformity.
10. Limited English proficiency (e.g. unable to obtain informed consent for surgery without a translator)
11. Ward of the State children

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Luhmann, MD, Principal Investigator — St. Louis Children's Hospital
Locations (1):
- Barnes Jewish Hospital and St. Louis Children Hospital / Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 7 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 13.5 [12 to 17] | 14.4 [13 to 18] | 13.9 [12 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 15
BMI [Mean (Full Range); unit: kg/m^2] | 22.8 [18.5 to 36] | 23.4 [19.9 to 30.5] | 23.1 [18.5 to 30.5]

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: measured in morphine-equivalent dosage (MED)
Time Frame: up to 6 weeks after surgery
Measure: Mean (Full Range); unit: Morphine ME
Groups:
- Study: Lidocaine: Will receive intravenous lidocaine during and after posterior spinal fusion for AIS
- Control: Control: Will receive saline placebo during and after surgery
Arm/Group | Study | Control
Number analyzed (Participants) | 8 | 7
Morphine ME | 63.7 [41.3 to 105.3] | 119.3 [38.1 to 180.1]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Study | Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT03893318/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT03893318/ICF_001.pdf